CLINICAL TRIAL: NCT00643669
Title: 24 Hour IOP Lowering Efficacy of AL-3789
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C-07-65
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-3789 (Experimental): AL-3789 Sterile Suspension, single depot administration of 0.8 mL in the study eye
  Interventions: Drug: AL-3789 Sterile Suspension
- No treatment (No Intervention): Fellow eye, as randomized

INTERVENTIONS:
Drug: AL-3789 Sterile Suspension — Single administration by anterior juxtascleral depot
  Arms: AL-3789

SUMMARY:
The objective of this study was to describe the intraocular pressure-lowering efficacy of AL-3789 over a 24-hour period in patients with open-angle glaucoma compared to an untreated control. Patients received one treatment of AL-3789. Twenty-eight days after treatment, IOP was measured every 4 hours, beginning at 8 AM for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma and treated for at least 30 days prior to Screening Visit with a topical prostaglandin analog as monotherapy.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pregnant, intend to become pregnant, breastfeeding.
* Difference in IOP greater than 3 mm Hg between eyes at Screening Visit.
* Any form of glaucoma other than open-angle glaucoma.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure (IOP) | Day 28, Up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Inglewood, Inglewood, California, United States